CLINICAL TRIAL: NCT00906022
Title: EXPAND Study - Self Expanding Nitinol Stent Versus PTA With Optional Bailout Stenting in Case of PTA Failure in Patients With Symptomatic Critical Limb Ischemia or Severe Intermittent Claudication. A Prospective, Multi-center, Randomized Clinical Trail With Follow-up Investigations at 1, 3, 6, and 12 Months.
Brief Title: Self Expanding Nitinol Stent Versus Percutaneous Transluminal Arterial Angioplasty (PTA) With Optional Bailout Stenting in Case of PTA Failure in Patients With Symptomatic Critical Limb Ischemia or Severe Intermittent Claudication (EXPAND)
Acronym: EXPAND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C0801
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Patients With Symptomatic Critical Limb Ischemia; Severe Intermittent Claudication
Keywords: Below the Knee; Infrapopliteal arteries; nitinol; limb ischemia; claudication; self-expanding stent; duplex; angiography
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Astron Pulsar Stent (Experimental): Device: Astron Pulsar Stent
  Interventions: Device: Astron Pulsar Stent
- PTA alone (Active Comparator): Device: Balloon angioplasty alone
  Interventions: Device: PTA alone

INTERVENTIONS:
Device: Astron Pulsar Stent — Stenting with Astron Pulsar
  Arms: Astron Pulsar Stent
Device: PTA alone — Balloon angioplasty alone
  Arms: PTA alone

SUMMARY:
The clinical investigation is a prospective, international, multi-centre, randomized (1:1) trial with follow up investigations at 1, 3, 6 and 12 months. Patients will be randomized either to treatment with stenting with the Astron Pulsar SE (4 or 5 mm diameter) stent or to PTA with optional bailout stenting in case of PTA failure.

The primary objective of this study is to show clinical improvement in the outcome of patients with symptomatic critical limb ischemia or severe intermittent claudication (Rutherford 3, 4, 5) treated with the Astron Pulsar SE (4 or 5 mm diameter) in comparison with PTA or optional bailout stenting in case of PTA failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50 years
2. Patient has signed the patient informed consent.
3. Patient is willing to adhere to the follow up time points and to follow the requirements during the study
4. Patient has symptomatic critical limb ischemia or severe intermittent claudication classified as Rutherford category 3, 4 or 5.
5. Stenotic (> 50%) or occlusive atherosclerotic disease of the infrapopliteal arteries below the radiographic level of the knee joint and above the level of the ankle (includes the peroneotibial trunk, anterior tibial artery, posterior tibial artery and peroneal artery, excludes the popliteal artery), as determined by pre-procedure intra-arterial DSA (preferred) or conventional angiography.
6. Target (study) lesion to be treated is a de novo lesion (lesion ≤ 190 mm length). NOTE: Multiple or diffused lesion treatment is allowed as long as total lesion length ≤ 190 mm)
7. Reference vessel diameter is between 2.5 and 4.0 mm.
8. Target vessel: It must be possible to follow the vessel run-off to the foot and/or the wound area. NOTE: Patients with incomplete or abnormal anatomical run-off are NOT excluded. Important is to see that the there is a run-off to the foot and/or wound area even if collaterals are involved.
9. Haemodynamically significant inflow stenoses of vessels above the knee were successfully treated before.
10. Lesions must be crossed successfully with a guide wire and guide wire must be within the true lumen of the distal vessel.

Notes:

* Target vessel has to be defined; Target vessel = vessel with target lesion to be treated
* Target vessel: Multiple or diffused lesions with total length > 190 mm => inclusion criteria are NOT fulfilled
* NON-target vessel(s): haemodynamically significant lesion can be treated according to investigator's discretion

Exclusion Criteria:

1. Patient refuses treatment.
2. Patient is legally, physically or mentally unable to give consent.
3. ABI / TBI measurement is impossible.
4. Target lesion is pre-treated.
5. Target lesion lies within or adjacent to an aneurysm.
6. Acute thrombus present in the target limb.
7. The reference vessel diameter is not suitable for available stent size (RVD < 2.5 and > 4.0 mm).
8. Length of lesion requires more than one treatment device (lesion length > 190 mm)
9. Hybrid technique (bypass surgery and peripheral intervention with PTA or stent during the same session) is not allowed. Note: Allowed is if the patient got a P1 or P3 bypass in a previous session and it is possible to treat a distal lesion through that bypass in a separate session. Time window between bypass surgery and planned intervention must be at least 30 days.
10. Life-expectancy less than 12 months at the time of screening.
11. Patient has a known allergy to heparin, aspirin, clopidogrel or other anticoagulant/ antiplatelet therapies, to nickel or contrast media or is unwilling to tolerate such therapies.
12. Patient has bleeding diatheses
13. Patient is currently enrolled in another investigational device or drug trial.
14. Patient took part in another investigational device or drug trial within 3 months prior to screening.
15. Patient is currently breast-feeding, pregnant or intends to become pregnant.
16. Myocardial infarction without coronary revascularization < 6 months prior to screening and with coronary revascularization < 1 month prior to screening.
17. Previous coronary or peripheral bypass surgery within 30 days prior to screening.
18. Patient had a calculated creatinine clearance < 30 ml/min within 30 days prior to screening.
19. Patient had a stroke or TIA within the last 6 months prior to screening.
20. Patient had a major amputation of the target limb (defined as above the ankle) at the time of screening

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate of sustained clinical improvement at 12 months follow up. Sustained clinical improvement is defined as: Upward shift of at least +1 (for Rutherford category 3) or +2 (for Rutherford categories 4 and 5) on the Rutherford scale. | 12 months

SECONDARY OUTCOMES:
MAE rate, amputation rate, mortality rate, Maximum Walking Distance and Pain Free Walking Distance, Quality of Life, Binary restenosis rate, technical and device success, hemodynamic outcome | 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gefässzentrum Berlin, Evangelisches Krankenhaus KEH, Berlin, Germany

REFERENCES:
- [Derived] Schulte KL, Pilger E, Schellong S, Tan KT, Baumann F, Langhoff R, Torsello G, Zeller T, Amendt K, Brodmann M; EXPAND Investigators. Primary Self-EXPANDing Nitinol Stenting vs Balloon Angioplasty With Optional Bailout Stenting for the Treatment of Infrapopliteal Artery Disease in Patients With Severe Intermittent Claudication or Critical Limb Ischemia (EXPAND Study). J Endovasc Ther. 2015 Oct;22(5):690-7. doi: 10.1177/1526602815598955. Epub 2015 Aug 5. PMID 26245919